CLINICAL TRIAL: NCT01675843
Title: Ovarian Stimulation and Intrauterine Insemination in Women With Polycystic Ovarian Syndrome
Acronym: OSIPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Gibreel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG/4/2010
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Infertility; Polycystic Ovarian Syndrome; Intrauterine Insemination
Keywords: Infertility; PCOS; IUI
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): controlled ovarian hyperstimulation (COH) and intrauterine insemination (IUI)
  Interventions: Procedure: Intrauterine insemination (IUI)
- Group B (No Intervention): Controlled ovarian hyperstimulation (COH)+ Timed Intercourse (TI)

INTERVENTIONS:
Procedure: Intrauterine insemination (IUI) — The male semen is obtained then processed by swim up technique and then introduced into the uterus by special catheter.
  Other Names: IUI
  Arms: Group A

SUMMARY:
The study null hypothethesis is: intrauterine insemination (IUI) does not improve pregnancy rates in women with polycystic ovary syndrome. Infertile women with pcos will receive gonadotropins for ovarian stimulation and then randomize to either IUI or timed intercourse (TI)

ELIGIBILITY:
Inclusion Criteria:

- women who failed to get pregnant after 6 ovulation induction cycles with clomiphene citrate (cc) alone, despite of being ovulating with cc, having patent Fallopian tubes as confirmed by hysterosalpingography and their partners had fertile semen parameters according to criteria of World Health Organization (WHO 2010)

Exclusion Criteria:

male factor infertility

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Live Birth Rate | 20 months

SECONDARY OUTCOMES:
Clinical pregnancy rate | 16 months

OTHER OUTCOMES:
multiple pregnancy rate | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gibreel, MD, Principal Investigator — Mansoura University
Locations (1):
- Fertility Care Unit, Al Mansurah, Eldakahlia, Egypt